CLINICAL TRIAL: NCT01382693
Title: Effects of Involvement in a Group-based Creative Expression Program on Psychotropic Drug Use in Persons With Dementia in Long-term Care: a Cluster-randomized Pilot Study
Brief Title: Effects of Involvement in a Group-based Creative Expression Program on Psychotropic Drug Use in Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Winona Houser, Medical Student, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 36459 EP
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Dementia
Keywords: Behavioral symptoms; Long-term care
MeSH Terms: conditions — Dementia; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TimeSlips group storytelling program (Experimental)
  Interventions: Behavioral: TimeSlips
- Standard care activity program (Active Comparator)
  Interventions: Behavioral: Standard care activity program

INTERVENTIONS:
Behavioral: TimeSlips — TimeSlips is a group-based creative storytelling program for people with dementia. The intervention will be held twice a week for six weeks, in hour-long sessions.
  Other Names: creative expression program; storytelling program
  Arms: TimeSlips group storytelling program
Behavioral: Standard care activity program — Standard-of-care activities for the study site's skilled-nursing dementia Special Care Units.
  Arms: Standard care activity program

SUMMARY:
This project, a small-scale pilot study, will attempt to determine if involvement in a group-based creative expression program may correlate with a reduction in use of psychotropic drugs for persons with dementia.

DETAILED DESCRIPTION:
The study site has two skilled-nursing dementia Special Care Units. One unit will serve as a control with residents receiving the standard care activity program. The other unit will receive the standard care activity program as well as the TimeSlips storytelling program (two hour-long sessions per week for six weeks). The behavioral symptoms and psychotropic drug usage for both cohorts will be studied for eight months, the first four months with no intervention and the last four months with or without the six-week TimeSlips intervention.

ELIGIBILITY:
Inclusion Criteria:

* residence in one of two dementia special-care skilled nursing units at the study site
* clinical diagnosis of dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Rates of psychotropic drug prescriptions for study participants. | eight months

SECONDARY OUTCOMES:
Mood and behavior patterns | eight months

CONTACTS AND LOCATIONS:
Overall Officials: Winona S Houser, BA, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center; Daniel R George, PhD, Study Director — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Landis Homes, Lititz, Pennsylvania, United States